CLINICAL TRIAL: NCT03395262
Title: An Examination of a Novel Weight Loss Formula on Anthropometry and Indices of Cardiovascular Disease Risk
Brief Title: An Examination of a Weight Loss Formula on Health
Acronym: NB14
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Richard B. Kreider, Executive Director, Human Clinical Research Facility, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2016-0829FX
Record Dates: First submitted 2017-12-18; First posted 2018-01-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2017-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Exercise; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active with caffeine (Experimental): Novel formula with caffeine
  Interventions: Dietary Supplement: Active with caffeine
- Active without caffeine (Active Comparator): Novel formula without caffeine
  Interventions: Dietary Supplement: Active without caffeine
- Placebo (Placebo Comparator): Dextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active with caffeine — Novel formula with caffeine
  Arms: Active with caffeine
Dietary Supplement: Active without caffeine — Novel formula without caffeine
  Arms: Active without caffeine
Dietary Supplement: Placebo — Dextrose placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to examine a novel weight loss formula with and without common stimulants on anthropometry and indices of cardiovascular disease risk.

DETAILED DESCRIPTION:
Obesity remains a problem for overall health and risk for cardiovascular disease worldwide. While dietary modification and increased levels of physical activity remain steadfast recommendations, alternative strategies related to supplementation remain an interest for the general populace and medical communities. A potential objection to the use of dietary supplements is that they often contain stimulants designed to increase metabolism. However, consumers and health practitioners alike are wary of such formulae; hence, the continued investigation of non-stimulant supplements is warranted. Therefore the aim of this study is to examine a novel weight loss formula with and without common stimulants on anthropometry and indices of cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 25 and 34.9

Exclusion Criteria:

* Recent history of weight change (+/- 10 lbs. within the past 3 months)
* Uncontrolled metabolic disorders
* Uncontrolled cardiovascular disorders
* Currently taking prescription medications (birth control is allowed)
* Currently taking dietary supplements for weight loss
* Pregnant or plan to become pregnant
* Have an intolerance to caffeine or other natural stimulants

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Body Composition - Weight | Measured every 4 weeks for 12 weeks
  Changes in body weight (kg) analyzed with related body composition variables via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Body Composition - Fat Mass | Measured every 4 weeks for 12 weeks
  Changes in fat mass (kg) analyzed with related body composition variables via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Body Composition - Body Fat Percent | Measured every 4 weeks for 12 weeks
  Changes in body fat (%) analyzed with related body composition variables via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).

SECONDARY OUTCOMES:
Body Composition - Lean Tissue Mass | Measured every 4 weeks for 12 weeks
  Change in lean tissue mass (kg) analyzed with related body composition outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Body Composition - Bone Mass | Measured every 4 weeks for 12 weeks
  Change in bone mass (g) analyzed with related body composition outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Body Composition - Fat Free Mass | Measured every 4 weeks for 12 weeks
  Changes in fat free mass (sum of lean tissue mass and bone mass expressed in kg) analyzed with related body composition variables via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Body Composition - Total Body Water | Measured every 4 weeks for 12 weeks
  Change in total body water (L and %) and analyzed with related body composition outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Resting Energy Expenditure - Caloric Expenditure | Measured every 4 weeks for 12 weeks
  Change in resting energy expenditure expressed in absolute (kcals/d) and relative terms (kcals/kg/day) and analyzed with related resting energy expenditure outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Resting Energy Expenditure - Respiratory Exchange Ratio | Measured every 4 weeks for 12 weeks
  Change in resting respiratory exchange ratio (RER) as an indicator of carbohydrate and fat oxidation analyzed with related resting energy expenditure outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Anthropometric Measures - Waist Circumference | Measured every 4 weeks for 12 weeks
  Change in waist circumference (cm) analyzed with related anthropometric outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Anthropometric Measures - Hip Circumference | Measured every 4 weeks for 12 weeks
  Change in hip circumference (cm) analyzed with related anthropometric outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Anthropometric Measures - Waist to Hip Ratio | Measured every 4 weeks for 12 weeks
  Change in the ratio of waist to hip (waist / hip circumference) analyzed with related anthropometric outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Anthropometric Measures - Body Mass Index | Measured every 4 weeks for 12 weeks
  Change in body mass index (kg of body mass / height in meters squared) analyzed with related anthropometric outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Dietary Energy Intake - Total Caloric Intake | Measured every 4 weeks for 12 weeks
  Change in caloric/energy intake (kcals/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Dietary Energy Intake - Carbohydrate | Measured every 4 weeks for 12 weeks
  Change in dietary carbohydrate intake (grams/day and grams/kg/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Dietary Energy Intake - Fat | Measured every 4 weeks for 12 weeks
  Change in dietary fat intake (grams/day and grams/kg/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Dietary Energy Intake - Protein | Measured every 4 weeks for 12 weeks
  Change in dietary protein intake (grams/day and grams/kg/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Resting Hemodynamics - Heart Rate | Measured every 4 weeks for 12 weeks
  Changes in resting heart rate (bpm) analyzed with related resting hemodynamic outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Resting Hemodynamics - Systolic Blood Pressure | Measured every 4 weeks for 12 weeks
  Changes in resting systolic blood pressure (mmHg) analyzed with related resting hemodynamic outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Resting Hemodynamics - Diastolic Blood Pressure | Measured every 4 weeks for 12 weeks
  Changes in resting diastolic blood pressure (mmHg) analyzed with related resting hemodynamic outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Glucose Homeostasis - Blood Glucose | Measured every 4 weeks for 12 weeks
  Change in blood glucose (mg/dl) analyzed with related glucose homeostasis blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Glucose Homeostasis - Fasting Insulin | Measured every 4 weeks for 12 weeks
  Change in fasting insulin (µIU/mL) analyzed with related glucose homeostasis blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Glucose Homeostasis - Homeostatic Model Assessment of Insulin Resistance | Measured every 4 weeks for 12 weeks
  Change in Homeostatic Model Assessment of Insulin Resistance (Fasting insulin x Fasting glucose / 405) analyzed with related glucose homeostasis blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Lipid Profile - Triglyderides | Measured every 4 weeks for 12 weeks
  Change in triglycerides (mg/dl) analyzed with related lipid profile blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Lipid Profile - Total Cholesterol | Measured every 4 weeks for 12 weeks
  Change in total cholesterol (mg/dl) analyzed with related lipid profile blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Lipid Profile - High Density Lipoproteins | Measured every 4 weeks for 12 weeks
  Change in high density lipoproteins (mg/dl) analyzed with related lipid profile blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Lipid Profile - Low Density Lipoproteins | Measured every 4 weeks for 12 weeks
  Change in low density lipoproteins (mg/dl) analyzed with related lipid profile blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Lipid Profile - Total Cholesterol to HDL Ratio | Measured every 4 weeks for 12 weeks
  Change in the ratio of total cholesterol to high density lipoproteins (HDL) analyzed with related lipid profile blood chemistry markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Creatinine | Measured every 4 weeks for 12 weeks
  Change in creatinine (mg/dl) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Blood Urea Nitrogen | Measured every 4 weeks for 12 weeks
  Change in blood urea nitrogen (mg/dl) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Blood Urea Nitrogen to Creatinine Ratio | Measured every 4 weeks for 12 weeks
  Change in the ratio of blood urea nitrogen (mg/dl) to creatinine (mg/dl) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Alkaline Phosphatase | Measured every 4 weeks for 12 weeks
  Change in alkaline phosphatase (IU/L) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Alanine Amino Transaminase | Measured every 4 weeks for 12 weeks
  Change in alanine amino transaminase (IU/L) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Aspartate Amino Transaminase | Measured every 4 weeks for 12 weeks
  Change in aspartate amino transaminase (IU/L) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Creatine Kinase | Measured every 4 weeks for 12 weeks
  Change in creatine kinase (IU/L) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Catabolic Markers - Lactate Dehydrogenase | Measured every 4 weeks for 12 weeks
  Change in lactate dehydrogenase (IU/L) analyzed with related blood chemistry catabolic markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - White Blood Cell Counts - White Blood Cells | Measured every 4 weeks for 12 weeks
  Change in white blood cells (K/uL) analyzed with related white blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - White Blood Cell Counts - Lymphocytes | Measured every 4 weeks for 12 weeks
  Change in lymphocytes (K/uL) analyzed with related white blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - White Blood Cell Counts - Mid-Range Count | Measured every 4 weeks for 12 weeks
  Change in mid-range count (K/uL) analyzed with related white blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - White Blood Cell Counts - Granulocyte | Measured every 4 weeks for 12 weeks
  Change in granulocyte count (K/uL) analyzed with related white blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Red Cells | Measured every 4 weeks for 12 weeks
  Change in red cell count (M/uL) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Hemoglobin | Measured every 4 weeks for 12 weeks
  Change in hemoglobin (g/dl) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Hematocrit | Measured every 4 weeks for 12 weeks
  Change in hematocrit (%) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Mean Corpuscular Volume | Measured every 4 weeks for 12 weeks
  Change in mean corpuscular volume (fL) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Mean Corpuscular Hemoglobin | Measured every 4 weeks for 12 weeks
  Change in mean corpuscular hemoglobin (pg/cell) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Mean Corpuscular Hemoglobin Concentration | Measured every 4 weeks for 12 weeks
  Change in mean corpuscular hemoglobin concentration (g/dl) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Red Cell Distribution Width | Measured every 4 weeks for 12 weeks
  Change in red cell distribution width (%) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Platelet Count | Measured every 4 weeks for 12 weeks
  Change in platelet count (x103/uL) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Red Blood Cell Counts - Mean Platelet Volume | Measured every 4 weeks for 12 weeks
  Change in mean platelet volume (fL) analyzed with related red blood cell count markers of health via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Blood Chemistry Markers of Health - Appetite Hormone - Leptin | Measured every 4 weeks for 12 weeks
  Change in leptin levels (ng/ml) analyzed via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
International Physical Activity Questionnaire (IPAQ) - Work Domain | Measured every 4 weeks for 12 weeks
  Change in IPAQ work domain (MET minutes/week) analyzed with related IPAQ outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
International Physical Activity Questionnaire (IPAQ) - Active Transportation Domain | Measured every 4 weeks for 12 weeks
  Change in IPAQ active transportation domain (MET minutes/week) analyzed with related IPAQ outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
International Physical Activity Questionnaire (IPAQ) - Domestic and Garden/Yard Work Domain | Measured every 4 weeks for 12 weeks
  Change in IPAQ domestic and garden/yard work domain (MET minutes/week) analyzed with related IPAQ outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
International Physical Activity Questionnaire (IPAQ) - Leisure-Time Domain | Measured every 4 weeks for 12 weeks
  Change in IPAQ leisure-time domain (MET minutes/week) analyzed with related IPAQ outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
International Physical Activity Questionnaire (IPAQ) - Total Physical Activity Score | Measured every 4 weeks for 12 weeks
  Change in IPAQ leisure time domain (Total physical activity MET-minutes/week = sum of Total Work + Total Transport + Total Domestic and Garden + Total Leisure-Time MET-minutes/week scores) analyzed with related IPAQ outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Satiety Questionnaire - Perceptions of Appetite | Measured every 4 weeks for 12 weeks
  Changes in perceptions of appetite assessed using using a 0 to 10 Likert scale (0 was none, 2.5 was low, 5 was moderate, and 7.5 was high, and 10 was severe) and analyzed with related satiety questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Satiety Questionnaire - Perceptions of Hunger | Measured every 4 weeks for 12 weeks
  Changes in perceptions of hunger assessed using using a 0 to 10 Likert scale (0 was none, 2.5 was low, 5 was moderate, and 7.5 was high, and 10 was severe) and analyzed with related satiety questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Satiety Questionnaire - Perceptions of Satisfaction with Food | Measured every 4 weeks for 12 weeks
  Changes in perceptions of satisfaction with food assessed using using a 0 to 10 Likert scale (0 was none, 2.5 was low, 5 was moderate, and 7.5 was high, and 10 was severe) and analyzed with related satiety questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Satiety Questionnaire - Perceptions of Feelings of Fullness | Measured every 4 weeks for 12 weeks
  Changes in perceptions of feelings of fullness assessed using using a 0 to 10 Likert scale (0 was none, 2.5 was low, 5 was moderate, and 7.5 was high, and 10 was severe) and analyzed with related satiety questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Satiety Questionnaire - Perceptions of Diet / Eating Satisfaction | Measured every 4 weeks for 12 weeks
  Changes in perceptions of diet / eating satisfaction assessed using using a 0 to 10 Likert scale (0 was none, 2.5 was low, 5 was moderate, and 7.5 was high, and 10 was severe) and analyzed with related satiety questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Sleep Quality Questionnaire - Sleep Duration | Measured every 4 weeks for 12 weeks
  Changes in average reported sleep duration over the prior 48 hours analyzed with related sleep quality questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Sleep Quality Questionnaire - Sleep Quality | Measured every 4 weeks for 12 weeks
  Changes in rating of sleep quality over the prior 48 hours analyzed with related sleep quality questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Sleep Quality Questionnaire - Enthusiasm | Measured every 4 weeks for 12 weeks
  Changes in rating of enthusiasm over the prior 48 hours analyzed with related sleep quality questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Sleep Quality Questionnaire - Sleep Disturbances | Measured every 4 weeks for 12 weeks
  Changes in rating of sleep disturbances over the prior 48 hours analyzed with related sleep quality questionnaire outcomes via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Dizziness | Measured every 4 weeks for 12 weeks
  Change in perceptions of dizziness using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Headache | Measured every 4 weeks for 12 weeks
  Change in perceptions of headache using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Tachycardia | Measured every 4 weeks for 12 weeks
  Change in perceptions of tachycardia using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Palpitations | Measured every 4 weeks for 12 weeks
  Change in perceptions of palpitations using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Dyspnea | Measured every 4 weeks for 12 weeks
  Change in perceptions of dyspnea using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Nervousness | Measured every 4 weeks for 12 weeks
  Change in perceptions of nervousness using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Blurred Vision | Measured every 4 weeks for 12 weeks
  Change in perceptions of blurred vision using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).
Perceptions of Side Effects - Other Side Effects | Measured every 4 weeks for 12 weeks
  Change in perceptions of other side effects using a Likert scale [0 (none), 1-4 (light), 5-6 (mild), 7-9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses and mean changes from baseline with 95% confidence intervals (CI's).

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Lab - Human Clinical Research Facility, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No